CLINICAL TRIAL: NCT06250413
Title: Lyophilized Capsulated Autological Fecal Microbial Transplant to Restore Gut Microbiome After Treatment With Antibiotics
Brief Title: Autoflor -Lyophilized Capsulated Autological FMT to Restore Gut Microbiome After Treatment With Antibiotics
Acronym: FMT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Helve (Other)
Collaborators: University of Helsinki (Other)
Responsible Party: Sponsor-Investigator, Otto Helve, Docent, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: HUS/2231/2023
Record Dates: First submitted 2024-01-18; First posted 2024-02-09 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Microbial Colonization; Antibiotic Side Effect
Keywords: FMT; lyophilized; antibiotics
MeSH Terms: conditions — Communicable Diseases | interventions — Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants will be given 4 capsules containing fecal matter (Capsule 1) after treatment with antibiotics on day 7. Intervention group will be given placebo (Capsules 2) on day 28.
  Interventions: Other: FMT; Other: Placebo; Drug: Amox Clav
- Control (Placebo Comparator): The participants will be given 4 placebo capsules (Capsule 2) after treatment with antibiotics on day 7.
  Control group will be given FMT capsules (Capsules 1) as "rescue therapy" on day 28.
  Interventions: Other: FMT; Other: Placebo; Drug: Amox Clav

INTERVENTIONS:
Other: FMT — Capsulated oral auto fecal microbiota transplant
Other: Placebo — Capsulated hot chocolate powder
Drug: Amox Clav — 5 day course of Amoxicillin Clavulanic acid given to all participants
  Other Names: Amorion comp

SUMMARY:
In this clinical trial, our aim is to assess the effect of auto-FMT (Fecal microbiome transplantation) on the intestinal microbiota, after a course of antibiotics.

30 healthy adults are recruited. All are given a five day course of amoxicillin-clavulanate. The subjects are double blinded and randomized to two groups. Group A is given autologous FMT (auto-FMT) on day 7 (two days after the end of the course of antibiotics) and Group B is given auto-FMT on day 28 (23 days after the end of the course of antibiotics).

DETAILED DESCRIPTION:
The use of antibiotics also has short- and long-term disadvantages for the individual. In trials with human adults, oral intake of antibiotics has been shown to markedly affect the intestinal microbiota, by reducing the diversity and altering the composition, as well as by spreading of antibiotic resistance genes (AR).

Freeze dried FMT products have long lasting stability of fecal microbiota useful for encapsulation. The amount of capsules needed to digest is also much lower compared to using fresh or frozen material.

Anticipating a 25% drop-out we will recruit 40 healthy adults between 18-40 years of age. Inflammation status of the participants at recruitment will be tested by taking blood samples. A 100-150g sample of the participants feces is obtained. The feces will be tested for potential harmful pathogens.

50g of collected stool is processed within 6 h of passage, diluted in 0.85% NaCl, homogenized using a mixer. The fecal suspension is filtered through sterilized metal sieves under biological safety cabinet. The suspension is then centrifuged. Supernatant is then decanted into new centrifuge tubes and centrifuged. The upper bacterial pellet is resuspended in isotonic sodium chloride with 10% trehalose. The suspension is stored at -80°C up to two weeks before being lyophilized. The solution is lyophilized in a Lyoquest plus Ae85C (Telstar, Tarrasa, Spain) for 44 h, and the resulting product is encapsulated in hypromellose capsules (sizes 0, Capsugel Enprotect, Cambridge, MA, USA) and stored at 4°C. The protocol is applied from previous studies with capsulated FMT. Each capsule contains approximately 0.35g lyophilized stool extract. O'boy hot chocolate powder is used as placebo.

The 30 participants are randomized and double blinded into two groups, each having 15 subjects. All participants will be given a 5-day (Day 1-5) course of Amoxicillin + Clavulanate 875/125 mg × 2.

Group A Intervention group. The participants will be given 4 capsules containing fecal matter (Capsule 1) after treatment with antibiotics on day 7.

Group B Control group. The participants will be given 4 placebo capsules (Capsule 2) after treatment with antibiotics on day 7.

Group B will be given FMT capsules (Capsules 1) as "rescue therapy" on day 28. Group A will be given placebo (Capsules 2) as described earlier.

The capsules (at timepoints 7 and 28 days) are administered under the supervision of the research team. The capsules are swallowed with juice. Participants are asked to be on a clear liquid diet for 8 h prior to the intervention. No solid food should be taken within two hours of digesting the capsules. Otherwise, no restrictions to the diet are considered necessary. During the visit the participants are interviewed and ensured that no signs of infection have occurred and that there have been no significant changes in bowel function.

Fecal samples will be collected from all participants weekly starting from day 6 for 7 weeks until day 48 (total 7 samples (3 vials/sample)). The study samples are stored in stool collection containers in the home freezer (-18°C) until collected by the study personnel and stored there after at -80°C. Calprotectin samples are stored in the refrigerator until collected by the study personnel.

The participants will fill in a questionnaire including questions of any abdominal symptoms, defecation frequency, stool consistence, abdominal pain, nausea and other used medication weekly until 7 weeks. Use of additional antibiotics during the follow-up period leads to drop-out. Participants complete a quality of life (HRQoL) survey at day 1 (the introduction of antibiotics), on day 7 when auto-FMT/placebo (first intervention) is performed, on day 28 (second intervention) and at the end of the follow-up period (day 48) (http://www.15d-instrument.net/15d/).

Participants with fever, watery diarrhea (> 3 loose stools in 24 hours), bloody stools, abdominal pain and cramping) are tested for C. difficile. In case of fever, the CRP level and complete blood count are controlled. Participants with bloody stools will be excluded from the study.

Blood samples will be taken on days 7, 9, 28 and 30. 5mL of blood is gathered (C-reactive protein, complete blood count, plasma).

ELIGIBILITY:
Inclusion Criteria:

-previously healthy

Exclusion Criteria:

* IBD (inflammatory bowel disease)
* celiac disease
* abdominal symptoms such as diarrhea or constipation necessitating medical therapy
* pregnancy and breastfeeding
* allergy towards antibiotics penicillins
* allergy towards soya.
* trehalose intolerance.
* travelling outside of European Union during the last 3 months
* use of antibiotics during the last 3 months
* use of probiotics during the previous 2 weeks or during the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility and safety; Number of participants with treatment-related adverse events such as; nausea, vomiting, signs of infection such as elevation of CRP after receiving the capsules, bloody stools | 2 months
  The feasibility and safety of the transplantation process using lyophilized auto-FMT. All adverse events are reported, CRP is taken from all patients at the day of the transplant and 2 day after. The participants answer to weekly online questionaires including questions of any abdominal symptoms, defecation frequency, stool consistence, abdominal pain, nausea and other used medication weekly until 7 weeks.
Taxonomic restoration of the gut microbiome at day 27. | 1 month
  Quantitative PCR will be used for quantitative microbiota profiling.

SECONDARY OUTCOMES:
The percentage of participants with restoration of intestinal microbiome. | 3 months
  The investigators observe especially the influence of auto-FMT towards successful restoration of bacteria from beneficial groups, including Lachnospiraceae (family), Ruminococcaceae (family), and Bacteroidetes (phylum).
Magnitude and duration of GI-symptoms | 3 months
  The investigators will use questionaires filled by the participants.
Impact of FMT given to placebo group on day 28 on gut microbiome on day 48 | 3 months
  Quantitative PCR will be used for quantitative microbiota profiling.

CONTACTS AND LOCATIONS:
Overall Officials: Otto Helve, Docent, Study Director — University of Helsinki
Locations (1):
- Helsinki University Hospital, Helsinki, Uusimaa, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jernberg C, Lofmark S, Edlund C, Jansson JK. Long-term impacts of antibiotic exposure on the human intestinal microbiota. Microbiology (Reading). 2010 Nov;156(Pt 11):3216-3223. doi: 10.1099/mic.0.040618-0. Epub 2010 Aug 12. PMID 20705661
- [Background] Reygner J, Charrueau C, Delannoy J, Mayeur C, Robert V, Cuinat C, Meylheuc T, Mauras A, Augustin J, Nicolis I, Modoux M, Joly F, Waligora-Dupriet AJ, Thomas M, Kapel N. Freeze-dried fecal samples are biologically active after long-lasting storage and suited to fecal microbiota transplantation in a preclinical murine model of Clostridioides difficile infection. Gut Microbes. 2020 Sep 2;11(5):1405-1422. doi: 10.1080/19490976.2020.1759489. Epub 2020 Jun 5. PMID 32501140
- [Result] Suez J, Zmora N, Zilberman-Schapira G, Mor U, Dori-Bachash M, Bashiardes S, Zur M, Regev-Lehavi D, Ben-Zeev Brik R, Federici S, Horn M, Cohen Y, Moor AE, Zeevi D, Korem T, Kotler E, Harmelin A, Itzkovitz S, Maharshak N, Shibolet O, Pevsner-Fischer M, Shapiro H, Sharon I, Halpern Z, Segal E, Elinav E. Post-Antibiotic Gut Mucosal Microbiome Reconstitution Is Impaired by Probiotics and Improved by Autologous FMT. Cell. 2018 Sep 6;174(6):1406-1423.e16. doi: 10.1016/j.cell.2018.08.047. PMID 30193113
- [Result] Bulow C, Langdon A, Hink T, Wallace M, Reske KA, Patel S, Sun X, Seiler S, Jones S, Kwon JH, Burnham CA, Dantas G, Dubberke ER. Impact of Amoxicillin-Clavulanate followed by Autologous Fecal Microbiota Transplantation on Fecal Microbiome Structure and Metabolic Potential. mSphere. 2018 Nov 21;3(6):e00588-18. doi: 10.1128/mSphereDirect.00588-18. PMID 30463925
- [Result] Taur Y, Coyte K, Schluter J, Robilotti E, Figueroa C, Gjonbalaj M, Littmann ER, Ling L, Miller L, Gyaltshen Y, Fontana E, Morjaria S, Gyurkocza B, Perales MA, Castro-Malaspina H, Tamari R, Ponce D, Koehne G, Barker J, Jakubowski A, Papadopoulos E, Dahi P, Sauter C, Shaffer B, Young JW, Peled J, Meagher RC, Jenq RR, van den Brink MRM, Giralt SA, Pamer EG, Xavier JB. Reconstitution of the gut microbiota of antibiotic-treated patients by autologous fecal microbiota transplant. Sci Transl Med. 2018 Sep 26;10(460):eaap9489. doi: 10.1126/scitranslmed.aap9489. PMID 30257956